CLINICAL TRIAL: NCT05714891
Title: Neoadjuvant Platform Trial in Patients With Surgically Resectable Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Neoadjuvant Platform Trial in Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I242
Record Dates: First submitted 2023-01-04; First posted 2023-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: NSCLC
MeSH Terms: interventions — JDQ443

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy (JDQ443) followed by surgery. (ARM CLOSED) (Experimental): If *MPR/cPR* - standard of care adjuvant treatment may be followed by experimental adjuvant therapy (JDQ443)
  *Major Pathological Response (MPR)/ Complete Pathological Response (cPR)
  Interventions: Drug: JDQ443

INTERVENTIONS:
Drug: JDQ443 — Dose will be assigned at enrollment

SUMMARY:
This study is being done to answer the following question: What are the effects of new treatments on non-small cell lung cancer before surgery?

DETAILED DESCRIPTION:
The purpose of the pre-study screening is to test for biomarkers. The testing will be done using a sample of your tumor tissue. Each substudy will be looking at what effects a new drug has on the patients and their lung cancer, as well as any side effects of the treatment. The purpose of each substudy is to see if the biomarkers that were identified at screening can be used to determine treatment outcomes, like how the cancer cells respond to treatment and whether the study drug will shrink the tumour before surgery and prevent it from returning after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of primary NSCLC within 90 days of enrollment to a substudy, according to WHO Classification of Tumours
* Unless otherwise specified in a substudy, patients must be classified as Stage IA2 to IIIA according to the AJCC 8th edition TNM classification with disease that is amenable to anatomical surgical resection.
* Pre-surgical staging of patients with newly diagnosed lung cancer should include: CT thorax, abdomen and pelvis; PET scan imaging; Brain MRI or CT brain with IV contrast. Patients with mediastinal lymph nodes suspicious for metastases on PET imaging are required to undergo invasive staging by EBUS or mediastinoscopy to confirm or disprove pathological involvement of suspected nodes.
* All patients must have evaluable disease as defined by RECIST 1.1 although measurable disease is recommended.
* Patients that are eligible for one or more substudies must consent for release of tissue biopsies, surgical specimens and blood samples for conduct of tissue analyses. If there is insufficient tissue to conduct the proposed research studies without exhausting the diagnostic biopsies, please consult CCTG
* Patients must be ≥ 18 years of age
* No prior anticancer therapy for treatment of NSCLC. Patients with a history of NSCLC treated in the curative setting may be eligible but must be discussed with CCTG prior to enrollment
* Patient must have an ECOG performance status of 0 or 1
* Patients with synchronous primary tumours may be eligible if all of the following conditions are met:

  * The synchronous tumour is located within the planned resection area
  * The radiological appearance of the tumour is compatible with ground-glass opacity (GGO)
  * The synchronous tumour is not FDG-avid on PET imaging
  * The local multidisciplinary thoracic oncology tumour board has approved the surgical treatment plan
* Surgery for participants enrolled on this protocol will be according to generally accepted standards of care. Operative approach (VATS, RATS vs open) will be determined by the surgeon. Accepted types of resection must aim to achieve an R0 resection, as defined by the IASLC, including the highest resected mediastinal being negative for carcinoma.
* Unless otherwise specified in specific substudies, surgery must be performed between 2 to 4 weeks following the last dose of neoadjuvant therapy
* Patients must have adequate organ and marrow function within 7 days prior to enrollment. Some substudies may require different cutoff values.
* Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements.
* Patient is able and willing to complete the Patient Related Outcomes questionnaire
* Patients must be accessible for treatment and follow-up.
* Protocol treatment is to begin within 2 working days of patient enrollment
* Women/men of childbearing potential must have agreed to use a highly effective contraceptive method

Exclusion Criteria:

* Presence of locally advanced, unresectable cancer (regardless of stage), or metastatic cancer (Stage IV).
* Patients with a history of other malignancy may be eligible if curatively treated and/or the malignancy does not affect the determination of safety or efficacy of the investigational regimen (must be confirmed with CCTG).
* Clinically significant, uncontrolled cardiac disease and/or recent cardiac events (within 6 months), such as:

  * Unstable angina or myocardial infarction within 6 months prior to enrollment;
  * Symptomatic congestive heart failure (defined as New York Heart Association Grade II or greater);,
  * Documented cardiomyopathy;,
  * Clinically significant cardiac arrhythmias; (Note: patients with clinically controlled, asymptomatic atrial arrhythmias without any ventricular function compromise may be eligible; please consult CCTG).
  * Uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, unless controlled prior to first dose of study treatment.
  * Patients with a significant cardiac history, even if controlled, should have LVEF ≥ 50%
* History or current diagnosis of ECG abnormalities indicating significant risk of safety for participants participating in the study such as:

  * Concomitant clinically significant cardiac arrhythmias e.g. sustained ventricular tachycardia, and clinically significant second or third-degree AV block without a pacemaker;
  * History of familial long QT syndrome or known family history of Torsades de Pointes;
  * Resting QT interval corrected with Fridericia's formula (QTcF) > 480 msec on screening ECG or congenital long QT syndrome.
* Patients with prior allogenic bone marrow transplant, double umbilical cord blood transplantation (dUCBT) or solid organ transplant.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol. This includes but is not limited to:

  * Known clinical diagnosis of tuberculosis;
  * Pneumonitis or any history of pneumonitis requiring steroids (any dose);
  * Known primary immunodeficiency;
  * For Hepatitis B (HBV), Hepatitis C (HCV) and human immunodeficiency virus (HIV) infections, requirements will be substudy dependent.
* History of hypersensitivity to any drugs in any substudy, or to drugs of similar chemical class.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.
* Pregnant or breastfeeding women.
* Patients who are unable to swallow oral medication and/or have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the specific substudy drug(s)
* Patients with a history of non-compliance to medical regimens.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Identify promising neoadjuvant treatment regimens for NSCLC for later validation in randomized clinical trials, by evaluating major pathological response rates (MPR) | 3 years

SECONDARY OUTCOMES:
Number and severity of adverse events as per CTCAE version 5.0 | 3 years
Overall response rate using RECIST 1.1 | 3 years
Pathological complete response rate (pCR) | 3 years
Event-free survival at 2 years | 3 years
Completeness of surgical resection using the Residual (R) Tumor Classification | 3 years
Access to surgery (rate of open, video-assisted and robotic-assisted thoracic surgery) | 3 years
Rate (and reasons) of surgical access conversion (from video-assisted or robotic-assisted thoracic surgery to open surgery) | 3 years
Extent of surgery (rate of surgery types: wedge resection, segmentectomy, lobectomy, completion lobectomy, sleeve lobectomy, bilobectomy, pneumonectomy, major airway resection, and other) | 3 years
Extent of perihilar/lobar fibrosis and mediastinal adhesions (as per the Lee et al. (JTO, 2021) grading scale) | 3 years
Tumour downstaging: rate of patients with post-surgical downstaging when comparing cTNM and pTNM | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Spicer, Study Chair — McGill University, Montreal, QC Canada; Normand Blais, Study Chair — CHUM-Centre Hospitalier de l'Universite de Montreal, QC Canada
Locations (8):
- Canada (8):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre Research Inc., London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University, Montreal, Quebec
  - University Institute of Cardiology and, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No